CLINICAL TRIAL: NCT00453830
Title: Laparoscopic Versus Open Sigmoid Colectomy for Diverticular Disease: A Prospective Randomized Single-Blind Trial
Brief Title: Laparoscopic Versus Open Sigmoid Colectomy for Diverticular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Pascal Gervaz, University Hospital Geneva
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CER 04-179
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Diverticulitis
Keywords: Diverticulitis; laparoscopy; short term outcome
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: laparoscopic sigmoid resection — a laparoscopic 5 trocars approach for left colon mobilization, sigmoid colon transsection and intracorporeal colorectal anastomosis
  Other Names: laparoscopic-assisted sigmoid resection

SUMMARY:
Aim: This is a prospective, randomized comparison of traditional open (OS) and laparoscopic sigmoidectomy (LS) in patients with complicated diverticular disease. The study is designed in order to minimize bias by standardizing the two procedures and blinding patients and nurses during the preoperative and early postoperative period.

Hypothesis: A laparoscopic approach for sigmoidectomy has significant advantages over the open technique with respect to postoperative pain, duration of ileus, length of hospital stay, and perioperative morbidity.

Methods: Patients with complicated diverticular disease who are candidates for elective sigmoidectomy will be randomized the day before surgery, and anaesthetic technique and postoperative management will be standardized between groups. Surgeons with experience in both laparoscopic-assisted and open colectomy will perform both types of procedures. At the end of the operation, identical, opaque wound dressings will be applied and left in place until postoperative day 4. Both patients and nursing staff will therefore be blinded to the type of surgical technique during the early postoperative period.

Endpoints:

A) Postoperative pain assessed by the Visual Analog Scale at postoperative days 1, 2, and 3.

B) Postoperative intake of systemic opiates (morphine)

C) Duration of postoperative ileus, quantified by the interval in hours between the end of the procedure and passage of first stool.

D) Duration of hospital stay.

E) Surgical complications, such as wound infection, anastomotic leakage, bleeding

F) General medical complications, such as cardiopulmonary, pneumonia, and renal failure.

Rationale: This study will determine whether a laparoscopic sigmoidectomy is associated with significant clinical advantages over the traditional open approach when patients with complicated diverticular disease are blinded to the operative technique.

DETAILED DESCRIPTION:
Colonic diverticulosis is an increasingly common condition in the Western societies; in our country, a third of the population is affected by the 6th decade and two-thirds by the 9th decade. Fortunately, a majority of patients with diverticulosis remain asymptomatic; diverticulitis, the most common presentation of complicated diverticular disease, has an estimated incidence of 10 patients per 100,000/year.

Colonic diverticular disease is usually restricted to the sigmoid colon, and conservative treatment with antibiotics is indicated in cases of a first attack of uncomplicated diverticulitis, the rationale being that a majority of patients treated for a first episode of acute inflammation will eventually recover and have no further problems.

Elective sigmoidectomy is currently recommended in the following clinical situations:

1. Patients who had two episodes of uncomplicated diverticulitis.
2. Patients who had one episode of complicated (perforated) diverticulitis, with either pericolic of pelvic abscesses (Hinchey stage I and II respectively), fistula formation and/or stenosis.

Resection of the sigmoid colon is now commonly performed by laparoscopy, and a number of non-randomized publications have demonstrated that this approach is safe and feasible in patients with diverticular disease. The theoretical advantages of celioscopy over the open techniques include decreased postoperative pain, a shorter duration of postoperative ileus and hospital stay, and improved cosmetic. Surprisingly, however, most published data on the topic are restricted to case-control series, and so far the putative advantages of laparoscopy have not been substantiated through a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diverticular disease of sigmoid colon documented by colonoscopy AND 2 episodes of uncomplicated diverticulitis, one at least being documented with CT scan OR 1 episode of complicated diverticulitis, i.e. perforation, with or without pericolic abscess or pelvic abscess requiring percutaneous drain

Exclusion Criteria:

* Age < 18
* Associated colon cancer or any condition requiring extended colectomy
* BMI > 35
* Emergency procedure
* Use of opiates and/or analgesics within 48 hours preceding the surgical procedure
* Patient unable to communicate in French, English or German
* Any cognitive impairment (psychiatric disorder, Alzheimer's disease, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain at days 1, 2 and 3 | 7 days
Morphine requirements at days 1, 2 and 3 | 4 days
Duration of postoperative ileus | 10 days

SECONDARY OUTCOMES:
Medical complications | 30 days
Surgical complications | 30 days
Duration of surgical procedure | 1 days
Duration of hospital stay | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Morel, MD, Study Chair — University Hospital Geneva - Department of Surgery
Locations (1):
- Department of Surgery, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Gervaz P, Mugnier-Konrad B, Morel P, Huber O, Inan I. Laparoscopic versus open sigmoid resection for diverticulitis: long-term results of a prospective, randomized trial. Surg Endosc. 2011 Oct;25(10):3373-8. doi: 10.1007/s00464-011-1728-8. Epub 2011 May 10. PMID 21556992
- [Derived] Gervaz P, Inan I, Perneger T, Schiffer E, Morel P. A prospective, randomized, single-blind comparison of laparoscopic versus open sigmoid colectomy for diverticulitis. Ann Surg. 2010 Jul;252(1):3-8. doi: 10.1097/SLA.0b013e3181dbb5a5. PMID 20505508